CLINICAL TRIAL: NCT05471934
Title: Satisfaction Survey - Cicaplast Mains
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: LRP14011-CICAPLAST BAUME B5
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Hand Eczema; Hand Dermatoses
MeSH Terms: conditions — Hand Dermatoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The participants presenting with hand problems and meeting the inclusion criteria are asked to apply the study product for one month. They are evaluated before and after treatment.

DETAILED DESCRIPTION:
The international, open, observational survey is conducted in 3 different countries.

Regarding the statistical analysis, the global satisfaction is described in 5 classes and in 2 classes "Satisfied + Very satisfied" vs. "Neither satisfied nor dissatisfied + Not so satisfied + Not at all satisfied". The 95% Confidence Interval (CI) of the percent of "Satisfied + Very satisfied" is also given.

On patients who already used cream at the inclusion, the following analyses are performed:

* Cross-tabulation between both visits,
* Test of the evolution between both visits using a special procedure for ordinal data with repeated measures,
* Description of a summary variable in 3 classes (Improved / No change / Worsened).

For the analysis of the hands problems, each sign is described at the inclusion and at the evaluation visit. The difference Evaluation-Inclusion is also given. The evolution of the sign is performed by a Wilcoxon test for matched samples.

ELIGIBILITY:
Inclusion Criteria:

* professionals that work on different activities related to hair in a beauty salon
* professionals presenting with current hand problems such as dryness, redness, irritations, cracks and fissures

Exclusion Criteria:

- professionals that do not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population corresponds to hairdressing professionals who are in permanent contact with irritating products (e.g. shampoos, hair colorants, oxidants, ...).
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
satisfaction rate | from baseline to Day28
  satisfaction questionnaire with a 5-point scale

SECONDARY OUTCOMES:
evaluation of hands problems (dryness, redness, irritations, cracks, fissures) | from baseline to Day28
  evaluation on a 10-point scale (0 Not at all to 10 Very strong)

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Kerob, Study Director — Cosmetique Active International
Locations (3):
- Dermatology practices, Roma, Italy
- Dermatology practices, Warsaw, Poland
- Dermatology practices, Ljubljana, Slovenia